CLINICAL TRIAL: NCT01553760
Title: The Use of an Anterior Chamber Maintainer as a Sole Fluid Source in Micro Incision Cataract Surgery as Compared to a Standard Phacoemulsification Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Abulafia Adi, MD, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 0163-11-MMC
Record Dates: First submitted 2012-02-19; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Cataract
Keywords: Cataract; TRI-MICS; ACM; MICS; phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tri-MICS (Experimental)
  Interventions: Procedure: Phacoemulsification using an ACM as the sole fluid source
- Conventional Phaco (Active Comparator)
  Interventions: Procedure: Conventional Phaco

INTERVENTIONS:
Procedure: Phacoemulsification using an ACM as the sole fluid source — A Tri-MICS system will be used with a sleeveless Kelman 20G tip through a 1.1mm CCI. A specialized 19G anterior chamber maintainer, with thin walls and a large internal diameter of 0.9mm will be inserted through a 1.1mm CCI.
  Arms: Tri-MICS
Procedure: Conventional Phaco — a conventional Phaco with sleeved Kelman 20G tip, through a 2.4mm CCI
  Arms: Conventional Phaco

SUMMARY:
The purpose of this study is to compare the use of an Anterior Chamber Maintainer (ACM) as the sole fluid source in phacoemulsification micro incision cataract surgery (using 1.1mm corneal incision) as opposed to conventional coaxial phacoemulsification (using 2.4mm corneal incision).

DETAILED DESCRIPTION:
Three-port Micro Incision Cataract Surgery (Tri-MICS) is a technique suggested by Professor Assia. The idea (principle) behind the Tri-MICS technique is the use of a sleeveless phaco needle which is introduced via a tiny incision (1.1mm). An additional corneal incision is made for the introduction of a second surgical instrument, and a third for an ACM as an exclusive source for the infusion - this saves the need for an additional instrument. The ACM that will be used in this study (AVI New York) is a small metal tube with an external diameter of 1.1 mm, and an internal diameter of 0.9 mm and was developed specifically for this use. This type of ACM has been used in hundreds of surgeries and has been found to be both effective and safe.

This procedure has 4 clear advantages:

1. The implementation of three corneal incisions, 1.1 mm wide with an angle of approximately 120 degrees between them - neutrality regarding astigmatism versus the Biaxial-MICS.
2. This procedure does not require any special medical instruments, for example; new phaco instruments which are specifically adapted for the MICS approach at the cost of tens of thousands of dollars.
3. This procedure allows a free use of the surgeon's second hand.
4. A fixed intraocular infusion keeps the intraocular pressure (IOP) and anterior chamber volume constant and stable.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral Cataract
* Ability to understand and sign on an inform consent form.
* whiling to undergo bilateral cataract surgery.

Exclusion Criteria:

* Mature Cataract
* PXF
* Uveitis
* Corneal Pathology
* Endothelial cell density<1500 cells/mm
* Glaucoma
* Extreme Hyperopia / shallow anterior chamber
* Extreme Myopia
* s/p Ophthalmic Trauma / Surgery
* Allergy to Penicillin / IOD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Corneal temperature | up to 12 months
  Continuous corneal temperature will be measured during cataract surgery using an infra red thermal imaging system

SECONDARY OUTCOMES:
Anterior chamber stability | up to 12 months
  Anterior chamber stability will be accessed during cataract surgery by the surgeon and post op by two different observers using surgery video record.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel